# A Physician-Initiated Multiple-Dose, Single Period, Phase 0-I Dose Ranging Study to Examine Levellor<sup>TM</sup> HypoSpray Human Insulin Adult Healthy Volunteer Patients

Protocol No.: LEV 101-D-022521

ClinicalTrials.gov Reference NCT04857320

# Criteria for evaluation: Statistical Analysis Plan

21st APRIL, 2021 Version 1.3

SPONSOR: Langford Research Institute

Principal Investigator: William D. Kirsh, D.O., M.P.H.



Approved by Langford Research Institutional Review Board April 21st, 2021

#### **AMENDMENTS:**

| 1. | 2. | 3. | 4. |
|----|----|----|----|

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable laws and regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you, which is indicated as privileged or confidential. Copyright 2020 Transdermal Delivery Solutions Corp dba HypoSpray Pharma.

| Criteria for |
|--------------|
| evaluation: |
| Statistical |
| Analysis |
| Plan |

### **Pharmacokinetics**

## Primary pharmacokinetic variables

The primary pharmacokinetic variables include: the reduction of serum glucose from baseline and at typical post prandial spikes and the amount of insulin necessary to accomplish this reduction.

In addition to 90% confidence intervals, the data will be summarized by medians, and maximum and minimum values.

The elimination half-life of Insulin will be compared using non-transformed data and parametric techniques.

Averages for the serum glucose and Post-prandial excursions will be compared against averages for experimental periods.